CLINICAL TRIAL: NCT06300593
Title: Evaluation of the Activity of Chronic Inflammation and Its Impact on Metabolic and Hormonal Parameters in Various PCOS Phenotypes
Brief Title: Activity of Chronic Inflammation in PCOS
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.292.2022-1
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS phenotypes; chronic inflammation; metabolic disorders; ovarian reserve
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PCOS phenotype A: clinical and/or biochemical hyperandrogenism (HA) + ovulatory dysfunction (OD) + polycystic ovarian morphology (PCOM)
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of C-reactive protein (CRP), interleukin-1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-alpha) in PCOS phenotypes A, B, C and D; Diagnostic Test: Evaluation of the correlation of serum concentrations of selected inflammatory markers (leucocytosis, CRP, IL-1, IL-6, IL-10, TNF-alpha) with metabolic and hormonal parameters
- PCOS phenotype B: HA + OD
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of C-reactive protein (CRP), interleukin-1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-alpha) in PCOS phenotypes A, B, C and D; Diagnostic Test: Evaluation of the correlation of serum concentrations of selected inflammatory markers (leucocytosis, CRP, IL-1, IL-6, IL-10, TNF-alpha) with metabolic and hormonal parameters
- PCOS phenotype C: HA + PCOM
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of C-reactive protein (CRP), interleukin-1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-alpha) in PCOS phenotypes A, B, C and D; Diagnostic Test: Evaluation of the correlation of serum concentrations of selected inflammatory markers (leucocytosis, CRP, IL-1, IL-6, IL-10, TNF-alpha) with metabolic and hormonal parameters
- PCOS phenotype D: OD + PCOM
  Interventions: Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of C-reactive protein (CRP), interleukin-1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-alpha) in PCOS phenotypes A, B, C and D; Diagnostic Test: Evaluation of the correlation of serum concentrations of selected inflammatory markers (leucocytosis, CRP, IL-1, IL-6, IL-10, TNF-alpha) with metabolic and hormonal parameters

INTERVENTIONS:
Diagnostic Test: Measurement and comparison of leucocytosis and concentrations of C-reactive protein (CRP), interleukin-1 (IL-1), IL-6, IL-10, Tumor Necrosis Factor (TNF-alpha) in PCOS phenotypes A, B, C and D — A venous blood sample of approximately 10 ml will be collected in the morning after 8 hours of fasting to determine and compare the above parameters of peripheral blood in the four study arms
Diagnostic Test: Evaluation of the correlation of serum concentrations of selected inflammatory markers (leucocytosis, CRP, IL-1, IL-6, IL-10, TNF-alpha) with metabolic and hormonal parameters — A venous blood sample of approximately 10 ml will be collected in the morning after 8 hours of fasting to test the above correlations in the four study arms

SUMMARY:
Chronic inflammation in polycystic ovary syndrome (PCOS) may be the result of dysregulation of cytokine production (due to insulin resistance, excess visceral fat and hyperandrogenemia), i.e., overproduction of pro-inflammatory factors (e.g. TNF, IL-1, IL-6) in relation to anti-inflammatory ones (IL-10). This condition may be an important link between obesity and insulin resistance, which is crucial in the etiopathogenesis of the syndrome. However, it is not known whether it results from the tendency to accumulate adipose tissue or is a feature of the syndrome itself. There is no data indicating the relationship between chronic inflammation and the severity of metabolic disorders and the value of ovarian reserve in women with various PCOS phenotypes.

DETAILED DESCRIPTION:
The study population will be characterized in terms of demographic (age, BMI), gynaecological (cycle length, menstrual pain, abnormal uterine bleeding) and obstetrics (pregnancies, childbirth, miscarriages) data. PCOS syndrome (and its phenotypes: A, B, C, D) will be recognized by the Rotterdam criteria. During hospitalization, blood samples will be collected for scheduled analyses (20 ml of blood in total).

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* PCOS syndrome confirmed by the Rotterdam criteria

Exclusion Criteria:

* absence of at least one ovary
* diagnosed and/or treated other metabolic disease
* diagnosed and/or treated other endocrine disease

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged 18-45, treated at the University Hospital in Krakow, diagnosed with PCOS confirmed by the Rotterdam criteria, phenotypes A, B, C, D, without other metabolic and endocrine diseases.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Values of inflammation parameters - leukocytosis in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of leukocyte count (n/µL) in peripheral blood in the four PCOS phenotypes
Values of inflammation parameters - C-reactive protein (CRP) in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of concentrations of CRP (mg/l) in peripheral blood in the four PCOS phenotypes
Values of inflammation parameters - IL-1 in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of concentrations of IL-1 (pg/ml) in peripheral blood in the four PCOS phenotypes
Values of inflammation parameters - IL-6 in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of concentrations of IL-6 (pg/ml) in peripheral blood in the four PCOS phenotypes
Values of inflammation parameters - IL-10 in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of concentrations of IL-10 (pg/ml) in peripheral blood in the four PCOS phenotypes
Values of inflammation parameters - TNF-alpha in peripheral blood in the four PCOS phenotypes | up to 3 months
  Measurement and comparison of concentrations of TNF-alpha (pg/ml) in peripheral blood in the four PCOS phenotypes

SECONDARY OUTCOMES:
Correlation between the HOMA-IR value and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the HOMA-IR value and inflammatory parameters: leukocyte count (n/µL)
Correlation between the homeostatic model assessment for insulin resistance (HOMA-IR) value and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the HOMA-IR value and inflammatory parameters: CRP (mg/l)
Correlation between the HOMA-IR value and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the HOMA-IR and inflammatory parameters: il-1 (pg/ml)
Correlation between the HOMA-IR value and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between HOMA-IR value and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of HOMA-IR and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the concentration of HOMA-IR and inflammatory parameters: il-10 (pg/ml)
Correlation between the HOMA-IR value and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the HOMA-IR value and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the body mass index (BMI) value and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the BMI value and inflammatory parameters: leukocyte count (n/µL)
Correlation between the BMI value and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the BMI value and inflammatory parameters: CRP (mg/l)
Correlation between the BMI value and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the BMI and inflammatory parameters: il-1 (pg/ml)
Correlation between the BMI value and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between BMI value and inflammatory parameters: il-6 (pg/ml)
Correlation between the concentration of BMI and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between BMI value and inflammatory parameters: il-10 (pg/ml)
Correlation between the BMI value and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between the BMI value and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of aspartate aminotransferase (AST) concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of AST concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: CRP (mg/l)
Correlation between the value of AST concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of AST concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of AST concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of AST concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AST concentration (U/l) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of alanine aminotransferase (ALT) concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of ALT concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: CRP (mg/l)
Correlation between the value of ALT concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of ALT concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of ALT concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of ALT concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between ALT concentration (U/l) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: CRP (mg/l)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of total bilirubin concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total bilirubin concentration (mg/dl) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: CRP (mg/l)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of total cholesterol concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between total cholesterol concentration (mg/dl) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of triglycerides concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of triglycerides concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: CRP (mg/l)
Correlation between the value of triglycerides concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of triglycerides concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of triglycerides concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of triglycerides concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between triglycerides concentration (mg/dl) and inflammatory parameters: TNF-alpha (pg/ml)
Correlation between the value of Anti-Müllerian hormone (AMH) concentration and the parameters of inflammation - leukocytosis in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: leukocyte count (n/µL)
Correlation between the value of AMH concentration and the parameters of inflammation - CRP in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: CRP (mg/l)
Correlation between the value of AMH concentration and the parameters of inflammation - il-1 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: il-1 (pg/ml)
Correlation between the value of AMH concentration and the parameters of inflammation - il-6 in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: il-6 (pg/ml)
Correlation between the value of AMH concentration and the parameters of inflammation - il-10 in in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: il-10 (pg/ml)
Correlation between the value of AMH concentration and the parameters of inflammation - TNF-alpha in the four PCOS phenotypes | up to 3 months
  Evaluation of the correlation between AMH concentration (pmol/l) and inflammatory parameters: TNF-alpha (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pitynski, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland